CLINICAL TRIAL: NCT02964832
Title: Assessment of Chest Compression Depth Obtained Using the Smartphone Application as an Educational Tool With New Attachment Device
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Joonbum Park, Assisstant professor of Emergency Medicine, Soonchunhyang University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: JPark1601
Record Dates: First submitted 2016-11-02; First posted 2016-11-16 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: Basic Cardiac Life Support
Keywords: Basic Cardiac Life Support, Education, Feedback

ARMS (3):
- PocketCPR;Grasp method (Active Comparator): Subject grasp a smartphone in the hand and compress the chest of manikin.
  Interventions: Device: Grasp method
- PocketCPR;Armband-in-hand method (Active Comparator): Grab the smartphone-contained-armband in hand when performing chest compression
  Interventions: Device: Armband-in-hand method
- PocketCPR;Armband-on-arm method (Active Comparator): Fix the smartphone-contained-armband on upperarm when performing chest compression
  Interventions: Device: Armband-on-arm method

INTERVENTIONS:
Device: Grasp method
  Arms: PocketCPR;Grasp method
Device: Armband-in-hand method
  Arms: PocketCPR;Armband-in-hand method
Device: Armband-on-arm method
  Arms: PocketCPR;Armband-on-arm method

SUMMARY:
To improve the quality of CPR education, we want to assess the validity and reliability of the feedback depth measured by smartphone applications according to the smartphone attachment sites as an educational tool. However, in the prior study, armband method showed overestimated chest compression depth. The reason of the overestimation was analyzed that the weight of the smartphone amplified the inertial force to produce additional linear movement. In this study, we will make new device to fix the smartphone on the arm and on the hand and compare the chest compression depth between CPR manikin and smartphone application.

ELIGIBILITY:
Inclusion Criteria:

* BLS provider or instructor

Exclusion Criteria:

* one who has physical problem in chest compression

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-03 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Assessment of validity of Chest compression depth by smartphone application,PocketCPR | Through study completion, average 4 weeks